CLINICAL TRIAL: NCT06131255
Title: ("The Role of the Glutamatergic Neurotransmission in Post- Partum Depression: an Integrated Molecular-pharmaco-imaging Study")
Brief Title: DRACULA1 Partum Depression: an Integrated Molecular-pharmaco-imaging Study")
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: DRACULA 1
Record Dates: First submitted 2023-04-13; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-03

CONDITIONS: Post-partum Depression
Keywords: post-partum depression; glutamatergic neurotransmission; antidepressants; citalopram
MeSH Terms: conditions — Depression, Postpartum | interventions — Citalopram

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Post-Partum Depression: 15 women with PPD referred to the S.C. Psychiatry of IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation and referred to the S.C. Neonatology and Neonatal Intensive Care Unit of the same institution for enrollment.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram — Patients will be administered citalopram, regardless of inclusion or non-inclusion in this study, on medical indication, as per normal clinical practice for disease management and according to the Summary of Product Characteristics (SPC). Patients will have two MRI scans done (at baseline and at 12 weeks after the start of therapy) to assess: brain volumetry, tissue amount of gray matter - GM - and white matter - WM

SUMMARY:
Post-partum depression (PPD) is a prevalent subtype of major depressive disorder that causes a significant distress to the woman and substantial impact on the whole family. Many studies implicate the glutamatergic system in pathological processes relevant to PPD disorders. There is evidence that cell adhesion molecules (CAMs) play a key role in how glutamatergic circuits wire up during development and how glutamatergic synapses, once formed, operate. However, it is unclear how dysregulation in diverse CAMs alter glutamatergic circuitries responsible for emotional and social behavior.

Here, the investigators propose to evaluate the molecular and neurobiological underpinnings of PPD focusing on CAMs at glutamatergic synapses by using an integrated approach from mouse models to human patients. Moreover, the investigators will also perform a pilot study to investigate the impact of selective antidepressants, known to be linked to CAMs, in both human and mice.

DETAILED DESCRIPTION:
Patients will be recruited by the physician in charge of the study or collaborators of the S.C. Neonatology and Neonatal Intensive Care Unit of the IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation upon referral from the S.C. Psychiatry of the same institution. In the study, exposure to citalopram treatment will be 12 weeks with follow-up every 4 weeks. At each participant, at the time of enrollment, will be assigned a unique code so that only the local investigators can trace the subject's identity. As part of a scheduled visit to assess the clinical diagnosis, the PPD patient will be offered to participate in the study, after the appropriate signing of informed consent, the verification of absence of criteria for exclusion and existence of the study inclusion criteria. If these criteria are met, some demographic and clinical medical history of the women with PPD will be collected, as already provided by clinical practice for the management of the disease. Patients will undergo MRI scanning at baseline at the S.C. Neuroradiology of the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico and will begin the pharmacological treatment with citalopram. It is emphasized that the administration of citalopram therapy for the treatment of depressive symptomatology will be proposed and carried out in the patient due to clinical needs, based on the judgment of the competent physician and as would already be the case in practice, thus completely independent of participation or non-participation in the present study. Neuroimaging data will be obtained with a Philips 3T magnetic resonance imaging MRI machine. For each patient enrolled in the study, a structural T1 sequence (3D MPRAGE) is acquired.

T1-weighted MRI images will be used to study the differences brain morphology, including the volumes of gray matter (GM) and white matter (WM) and voxel-based morphometry. In a comparison parallel between regions of interest (ROIs), regional volumes will be estimated using the automated anatomical labeling atlas (AAL) as a reference, with emphasis on the dorsolateral PFC (DL)/ventrolateral (VL), cingulate cortex, amygdala and hippocampus. Further regional analysis will allow estimation, in addition to cortical volumes and subcortical volumes, cortical thickness, cortical surface area, and the cortical gyrification of the Desikan-Killiany atlas regions. During treatment with citalopram, patients will be visited, as per standard clinical practice, every 4 weeks. At each of these follow-up visits will be administered to patients by medical specialists the Brief Psychiatric Rating Scale (BPRS) and the Hamilton Depression Rating Scale (HAM- D) to study symptomatology depression. Patients will be, instead, self-administered in Italian language the Maternal Postnatal Attachment Scale (MPAS) and the Parental Stress Index (PSI) to investigate mother-child attachment and parental stress. The time scheduled for completion of both scales will be about 40 minutes. At 12 weeks, as per practice, the MRI scan will be repeated at the S.C. Neuroradiology Department of the Foundation. The following variables will be collected as part of this study: socio-demographic variables (age, schooling, socio-economic);

* clinical/anamnestic variables (age of onset, duration of untreated treated, drug therapy, comorbidities, familiarity, substance abuse/dependence);
* BPRS and HAM-D scales scores for symptomatology assessment (T0, T1, T2, T3);
* MPAS and PSI scales scores for the assessment of mothers child attachment. (T0, T1, T2, T3);
* MRI scan data (T0, T3): the images will be used to study brain morphological differences, including GM and WM volumes, and voxel-based morphometry. In a parallel comparison between regions of interest (ROI), regional volumes will be estimated using as a reference the automated anatomical labeling atlas (AAL), with particular attention to the dorsolateral (DL)/ventrolateral (VL) PFC, cingulate cortex, amygdala and hippocampus. A further regional analysis will make it possible to estimate, in addition to cortical and subcortical volumes, the thickness cortical, cortical surface area and cortical gyrification of the Desikan-Killiany atlas regions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years;
* female gender;
* PPD diagnosed by DSM-5 structured clinical interview support (SCID-5) by trained medical personnel;
* comorbidity with metabolic syndrome, which can lead to brain damage and cognitive flaws;
* need to start citalopram therapy for clinical needs (and therefore independent of study participation) or already on therapy for no more than two weeks;
* moderate to severe depression according to the 17-item HAM-D (score 14-24);
* absence of disabling medical and/or neurological conditions, including heart attacks, brain injuries, neurodegenerative diseases, head trauma with loss of consciousness for more than 30 minutes;
* Absence of concomitant psychiatric therapies (antidepressants, antipsychotics of the first and second generation and mood stabilizers);
* absence of contraindications for MRI scanning;
* patients who have signed informed consent.

Exclusion Criteria:

* age below 18 years or above 40 years;
* diagnosis different from PPD based on SCID-5;
* absence of metabolic syndrome;
* low depression according to the 17-item HAM-D (score less than 14);
* presence of disabling medical and/or neurological conditions, including heart attacks, brain injuries, neurodegenerative diseases, head trauma with loss of consciousness for more than 30 minutes;
* presence of concomitant drug therapies (antidepressants, first- and second-generation antipsychotics and mood stabilizers);
* presence of contraindications for MRI scanning;
* presence of contraindications for citalopram;
* patients who have not signed informed consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Study Population: Women, aged 18 years to 40 years of age or older, with PPD who will be enrolled by the S.C. Neonatology and Neonatal Intensive Care Unit of the IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation upon referral from the S.C. Psychiatry of the same institution.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the citalopram effect on white matter morphology | 12 weeks
  Any statistically significant changes in brain volumetry and in the tissue amount of white matter (WM) will be evaluated after 12 weeks of treatment with citalopram.
Evaluate the citalopram effect on gray matter morphology | 12 weeks
  Any statistically significant changes in brain volumetry and in the tissue amount of gray matter (GM) will be evaluated after 12 weeks of treatment with citalopram.

SECONDARY OUTCOMES:
To evaluate the efficacy of citalopram on the clinical symptomatology of the PPD patients through the use of clinical scales | 12 weeks
  Variation of the score of HAM-D for measuring patients' symptomatology after 12 weeks after the start of treatment. Patients will be considered responsive if they have at least a 30% reduction from baseline HAM-D baseline after 12 weeks of treatment with citalopram.

OTHER OUTCOMES:
Assess the tolerability profile of the drug in the same patients | 12 weeks
  Evaluation of the serious and nonserious adverse events number judged by the medical staff to be related to the drug under study.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asahina H, Masuba A, Hirano S, Yuri K. Distribution of protocadherin 9 protein in the developing mouse nervous system. Neuroscience. 2012 Dec 6;225:88-104. doi: 10.1016/j.neuroscience.2012.09.006. Epub 2012 Sep 11. PMID 22982106
- [Background] Bambico FR, Belzung C. Novel insights into depression and antidepressants: a synergy between synaptogenesis and neurogenesis? Curr Top Behav Neurosci. 2013;15:243-91. doi: 10.1007/7854_2012_234. PMID 23271325
- [Background] Boku S, Nakagawa S, Toda H, Hishimoto A. Neural basis of major depressive disorder: Beyond monoamine hypothesis. Psychiatry Clin Neurosci. 2018 Jan;72(1):3-12. doi: 10.1111/pcn.12604. Epub 2017 Oct 19. PMID 28926161
- [Background] Bruining H, Matsui A, Oguro-Ando A, Kahn RS, Van't Spijker HM, Akkermans G, Stiedl O, van Engeland H, Koopmans B, van Lith HA, Oppelaar H, Tieland L, Nonkes LJ, Yagi T, Kaneko R, Burbach JP, Yamamoto N, Kas MJ. Genetic Mapping in Mice Reveals the Involvement of Pcdh9 in Long-Term Social and Object Recognition and Sensorimotor Development. Biol Psychiatry. 2015 Oct 1;78(7):485-95. doi: 10.1016/j.biopsych.2015.01.017. Epub 2015 Feb 7. PMID 25802080
- [Background] Cingolani LA, Thalhammer A, Yu LM, Catalano M, Ramos T, Colicos MA, Goda Y. Activity-dependent regulation of synaptic AMPA receptor composition and abundance by beta3 integrins. Neuron. 2008 Jun 12;58(5):749-62. doi: 10.1016/j.neuron.2008.04.011. PMID 18549786
- [Background] Davis AD, Hassel S, Arnott SR, Harris J, Lam RW, Milev R, Rotzinger S, Zamyadi M, Frey BN, Minuzzi L, Strother SC, MacQueen GM, Kennedy SH, Hall GB. White Matter Indices of Medication Response in Major Depression: A Diffusion Tensor Imaging Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Oct;4(10):913-924. doi: 10.1016/j.bpsc.2019.05.016. Epub 2019 Jun 12. PMID 31471185
- [Background] Postpartum Depression: Action Towards Causes and Treatment (PACT) Consortium. Heterogeneity of postpartum depression: a latent class analysis. Lancet Psychiatry. 2015 Jan;2(1):59-67. doi: 10.1016/S2215-0366(14)00055-8. Epub 2015 Jan 8. PMID 26359613
- [Background] Duric V, Banasr M, Stockmeier CA, Simen AA, Newton SS, Overholser JC, Jurjus GJ, Dieter L, Duman RS. Altered expression of synapse and glutamate related genes in post-mortem hippocampus of depressed subjects. Int J Neuropsychopharmacol. 2013 Feb;16(1):69-82. doi: 10.1017/S1461145712000016. Epub 2012 Feb 17. PMID 22339950